CLINICAL TRIAL: NCT01522950
Title: A Double-blind, Placebo-controlled, Randomized Study Examining the Effects of Nebivolol Compared to Atenolol on Endothelial Function and Cardiovascular Risk in Patients With Early Vascular Disease
Brief Title: A Study Examining the Effects of Nebivolol Compared to Atenolol on Endothelial Function
Acronym: EVIDENCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV-2014-20226
Record Dates: First submitted 2012-01-17; First posted 2012-02-01 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Hypertension
Keywords: hypertension; prevention; endothelial function
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Atenolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nebivolol (Active Comparator): 5 mg, continue for 1 month; dose titration to 10 mg, continue for 8 months. Dose may be returned to initiation levels if side effects occur.
  Interventions: Drug: Nebivolol
- Atenolol (Active Comparator): 25 mg, continue for 1 month; dose titration to 50 mg, continue for 8 months. Dose may be returned to initiation levels if side effects occur.
  Interventions: Drug: atenolol
- Placebo (Placebo Comparator): Continue for 1 month; dose titration to "high dose" placebo, continue for 8 months. Dose may be returned to initiation levels if side effects occur.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Nebivolol — 5 mg daily or 10 mg daily
  Arms: Nebivolol
Drug: atenolol — 25 mg daily or 50 mg daily
  Arms: Atenolol
Drug: placebo — one tablet daily
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study comparing the efficacy of nebivolol and atenolol at improving small artery elasticity and reducing cardiovascular disease risk in subjects with early vascular disease. Approximately 75 subjects with borderline/elevated blood pressures and impaired endothelial function, as measured by arterial elasticity scores, will be recruited and assigned to treatment groups using a block randomization scheme. Patients will be randomly allocated to nebivolol, atenolol or placebo, and then followed for 9 months.

DETAILED DESCRIPTION:
The Rasmussen Disease Score (RDS) test panel is the chosen methodology for this study. The 10 parameters of the RDS were selected because of their ability to quantify early structural and functional abnormalities in the vasculature and left ventricle which appear long before cardiovascular disease is present.

The RDS tests include: large and small artery elasticity (measured by pulse contour analysis), resting blood pressure, mild treadmill exercise test, carotid IMT, left ventricle mass, ECG, retinal vasculature evaluation, as well as quantification of serum NT-proBNP, and microalbuminuria. Quantitative results from these tests are converted into categorical classifications based on values stratified by age and gender when appropriate. The categorical data is scored as follows: normal = 0 points, borderline = 1 point, abnormal = 2 points. Point values from all parameters are summed to create the RDS, with values ranging from 0-20. Scores of 0-2 are classified as normal, 3-5 as early disease, and 6+ as advanced disease. Previous research has shown that the RDS is a powerful predictor of future cardiovascular events.

The small artery elasticity (C2) parameter is of particular interest as it is responsive to changes in NO levels and is an effective and reliable predictor of future hypertension and other cardiovascular events. Changes in C2 will serve as the primary outcome of this study. Similar studies using anti-hypertensive or lipid-lowering interventions have found significant improvements in C2 values.

Brachial artery flow-mediated dilation (FMD) measurements will also be measured as an index of endothelial function, although this method appears to be less sensitive to functional changes related to NO bioavailability than C2. Utilizing both FMD and C2 will allow comparison with previous studies and take advantage of a large sample size to further examine the relative sensitivity of each method for reliably measuring endothelial dysfunction.

The duration of intervention for this study is 9 months which is the minimum time to adequately detect improvement in left ventricle (LV) mass values. LV mass measurements are a critical component of a comprehensive assessment of cardiovascular health and have improved within this temporal window as a result of anti-hypertensive intervention.

ELIGIBILITY:
Inclusion Criteria:

* borderline blood pressure (120-145/80-90 mm Hg);
* borderline or abnormal small artery elasticity (C2) as measured by pulse contour analysis;
* treatment-naive for all blood pressure medications including diuretics for at least 30 days prior to baseline visit;
* able to walk on a treadmill for 3 minutes;
* female patients with reproductive potential must use an approved contraceptive method if appropriate (for example, intrauterine device [IUD], birth control pills, or barrier device during and for 1 month after the last dose of study drug;
* voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* history of intolerance to beta-blockers or clear contraindications to their use; current pharmaceutical treatment of blood pressure;
* known history of cardiovascular disease (myocardial infarction, coronary artery bypass graft, unstable angina, uncontrolled arrhythmias, stroke, etc.);
* known history of diabetes; known history of hepatic, renal or gastrointestinal disorder;
* known history of any illness that may cause additional risk (as determined by study investigator);
* pregnant or lactating women [when used during pregnancy, beta-blockers may cause fetal harm];
* participation in a concomitant clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay N Cohn, MD, Principal Investigator — University of Minnesota Medical Center
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Duprez DA, Florea N, Duval S, Koukol C, Cohn JN. Effect of nebivolol or atenolol vs. placebo on cardiovascular health in subjects with borderline blood pressure: the EVIDENCE study. J Hum Hypertens. 2017 Dec;32(1):20-25. doi: 10.1038/s41371-017-0019-9. Epub 2017 Nov 28. PMID 29184167

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nebivolol | Atenolol | Placebo
Started | 26 | 23 | 27
Completed | 20 | 18 | 22
Not Completed | 6 | 5 | 5
Not completed — Withdrawal by Subject | 3 | 2 | 1
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Death | 0 | 1 | 1
Not completed — Study Medication Sensitivity | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Atenolol | Placebo | Total
Number analyzed (Participants) | 20 | 18 | 22 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 16 | 16 | 50
  >=65 years | 2 | 2 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (14.5) | 50.8 (14) | 54 (9) | 50.7 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13 | 26
  Male | 11 | 14 | 9 | 34
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 22 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Small Artery Elasticity
Description: Change in small artery elasticity (a marker for endothelial function) from baseline to 9 months after intervention initiation.
Time Frame: baseline, 9 months
Measure: Mean (Standard Deviation); unit: (ml/mmHg × 100)
Arm/Group | Nebivolol | Atenolol | Placebo
Number analyzed (Participants) | 20 | 18 | 22
(ml/mmHg × 100) | 2.4 (2.1) | 1.0 (2.1) | 0.4 (1.7)

2. Secondary Outcome: Change in Large Artery Elasticity
Description: Change in large artery elasticity (a marker for endothelial function) from baseline to 9 months after intervention initiation.
Time Frame: baseline, 9 months
Measure: Mean (Standard Deviation); unit: (ml/mmHg × 10)
Arm/Group | Nebivolol | Atenolol | Placebo
Number analyzed (Participants) | 20 | 18 | 22
(ml/mmHg × 10) | 3.2 (5.4) | 2.9 (3.4) | 0.2 (2.6)

3. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure as measured by sphygmomanometer from baseline to 9 months after intervention initiation.
Time Frame: baseline, 9 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Atenolol | Placebo
Number analyzed (Participants) | 20 | 18 | 22
mmHg | -9 (12.9) | -13 (10.6) | -3.2 (12.4)

4. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure as measured by sphygmomanometer from baseline to 9 months after intervention initiation.
Time Frame: baseline, 9 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Atenolol | Placebo
Number analyzed (Participants) | 20 | 18 | 22
mmHg | -8.5 (10.1) | -8.5 (8.9) | -2.9 (6.7)

ADVERSE EVENTS:
Arm/Group | Nebivolol | Atenolol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/18 | 1/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 6/20 | 4/18 | 7/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol (N=20) | Atenolol (N=18) | Placebo (N=22)
Fatigue (General disorders) | 5 | 2 | 2
Headache (General disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 1
Dizziness (General disorders) | 0 | 0 | 1
Pruritus (General disorders) | 0 | 0 | 1
Hypertension (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT01522950/Prot_SAP_000.pdf